CLINICAL TRIAL: NCT06151301
Title: Evaluation of the Role of Poisoning Severity Score, Serum Procalcitonin and C-reactive Protein in Acute Hydrocarbon Intoxicated Cases Admitted to the Poison Control Center Ain Shams University Hospitals
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mera Gergis khalil, assistant lecteurer Forensic medicine and Toxicology department sohag univerisity hospital, Sohag University
Other Study IDs: Soh-Med-23-11-01MD
Record Dates: First submitted 2023-11-21; First posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Acute Hydrocarbon Toxicity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group: 20 subjects of apparently healthy persons for estimating the standard levels of the tested biomarkers.
  Interventions: Diagnostic Test: serum procalcitonin; Diagnostic Test: C-reactive protein
- case group: 60 patients divided into mild, moderate and severe toxicity according to the poisoning severity score.
  Interventions: Diagnostic Test: serum procalcitonin; Diagnostic Test: C-reactive protein

INTERVENTIONS:
Diagnostic Test: serum procalcitonin — predicting the severity of intoxication
Diagnostic Test: C-reactive protein — predicting the severity of intoxication

SUMMARY:
Hydrocarbons are a primary energy source in modern society. They are present in many common household and occupational products, including motor fuels, paint thinners, cleaning agents, lotions, and industrial solvents. Unfortunately, these products are also used as agents of abuse and typically inhaled .

They are derived mainly from petroleum (kerosene, gas, naphtha) or wood (turpentine, pine oil). They can be found in liquid, gas, or solid form depending on their properties. All hydrocarbons can be toxic, but aromatic (ring-shaped) and halogenated hydrocarbons typically have more severe toxicity .

Toxicity occurs in various ways including through inhalation, ingestion, aspiration, and dermal exposure. Frequently, these exposures occur during attempted recreational use of the substances and sometimes for self-injurious behavior

ELIGIBILITY:
Inclusion Criteria:

Patients of both sexes admitted to the Poison control center, Ain Shams university hospitals with acute hydrocarbon toxicity during the duration from December 2023 till December 2024 with a maximum number of 60 cases within 24 hours of intoxication.

Exclusion Criteria:

Patients with these criteria will be excluded:

* Cases > 24 hours of intoxication.
* Cases with occupational exposure to hydrocarbons.
* Pregnant females.
* Any cases received any treatment before arrival to the PCC.
* Cases suffering from cardiac, respiratory, renal, hepatic or haematological disorders.
* Cases presenting with fever.
* Cases with other causes that can increase levels of CRP & pro-calcitonin as bacterial infection, recent major trauma, major burn ,septic shock and medullary thyroid cancer.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of both sexes admitted to the Poison control center, Ain Shams university hospitals with acute hydrocarbon toxicity during the duration from December 2023 till December 2024 with a maximum number of 60 cases within 24 hours of intoxication
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Serum procalcitonin level | 1 year
  measuring the level of serum procalcitonin (reference range 0-0.05µg/L)

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams university Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No